CLINICAL TRIAL: NCT07052656
Title: Risk Factors and Outcomes in Patients Treated in Neurocritical Care
Acronym: EpiNIC
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Linn Hallqvist, MD, PhD, Consultant, Principal Investigator, Karolinska Institutet
Other Study IDs: K2022-6426; KI: 4-1998/2022 (Other: Karolinska Institutet)
Record Dates: First submitted 2025-05-28; First posted 2025-07-04 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Neuro-intensive Care Unit Patients; Subarachnoid Hemorrhage, Aneurysmal; Ischemic Stroke; Intracerebral Hemorrhage; Stroke, Acute; Meningitis; Epilepsy; Traumatic Brain Injury; Acute Brain Injuries; Acute Neurological Injury
MeSH Terms: conditions — Subarachnoid Hemorrhage; Ischemic Stroke; Cerebral Hemorrhage; Stroke; Meningitis; Epilepsy; Brain Injuries, Traumatic; Brain Injuries | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neuro-intensive care patients
  Interventions: Other: Observational study, participants are not assigned an intervention as part of the study.; Other: Transport modality

INTERVENTIONS:
Other: Observational study, participants are not assigned an intervention as part of the study. — Observational study, participants are not assigned an intervention as part of the study.
Other: Transport modality — Transfer modality to tertiary centers

SUMMARY:
The overall purpose of this epidemiologic research project is to provide a comprehensive exploration and analysis of critical elements within the neuro-intensive care process in Sweden. All aspects of intensive care management in critically ill patients with acute brain injury will be addressed. The analyses include description of patient characteristics, intensive care data, management and treatments, various aspects of short and long-term follow-up, mortality, regional- and sex-related differences. The long-term goal is to develop neuro-intensive care and management, to minimize in-hospital insults and secondary injuries, to improve diagnostics and follow-up, in order to reduce prolonged neurologic deficits and mortality in these patients.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission 2010 to 2024
* Clinical diagnosis of subarachnoid hemorrhage, intracranial hemorrhage or ischemic brain injury, traumatic brain injury, epilepsy, meningitis, encefalititis or other brain injury diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients 18 years or older treated in an ICU in Sweden with a clinical diagnosis of subarachnoid hemorrhage, intracranial hemorrhage, ischemic brain injury, traumatic brain injury, epilepsy, meningitis, encefalitis or other brain injury diagnosis from 2010 to 2024.
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Up to two years
  Mortality

SECONDARY OUTCOMES:
Morbidity | Up to two years
  Neuropsychiatric diagnoses, depression/anxiety), longterm sick leave, loss of income as a proxy for quality of life

OTHER OUTCOMES:
DAOH90 | 90 days
  Days alive and out of hospital
Complications | 90 days
  Rebleeding, secondary insults, cerebral infarctions

CONTACTS AND LOCATIONS:
Overall Officials: Linn Hallqvist, MD, PhD, Principal Investigator — Dep of Perioperative Medicine and Intensive care, Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided